CLINICAL TRIAL: NCT06397690
Title: UNCPM 22325 - Supporting Oral and Long-acting Pre-exposure Prophylaxis Decision Making Among Pregnant Women in Lilongwe, Malawi: a Feasibility Pilot Study
Brief Title: Supporting Oral and Long-acting PrEP Decision Making Among Pregnant Women in Lilongwe, Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0511; P30AI050410 (NIH)
Record Dates: First submitted 2024-04-19; First posted 2024-05-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: HIV Prevention
Keywords: PrEP in pregnancy and breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Choice for HIV Prevention (MyChoice) (Experimental): The MyChoice intervention consists of PrEP shared decision-making counseling delivered by a trained counselor. It begins with a review of HIV risk in pregnancy/breastfeeding including discussion of population-specific risk factors which may apply to the participant. Next, the counselor presents HIV prevention options including CAB-LA, daily oral PrEP, and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (product attributes and personal and interpersonal implications of each method). The counselor reviews information about these valued features for each offered method. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s).
  Interventions: Behavioral: My Choice for HIV Prevention (MyChoice)
- Standard of care (control arm) (Active Comparator): Participants randomized to the control arm will receive PrEP counseling as based on the current standard of care (SOC). The SOC counseling will be delivered by a trained study staff member. The SOC counselor PrEP counseling according to national guidelines. Control arm participants will receive comprehensive education on both the advantages and limitations of each PrEP method, including guidance on potential side effects. The SOC counselor will assess the woman's eligibility, willingness, and readiness to start using PrEP.
  Interventions: Behavioral: Standard of care (control arm)

INTERVENTIONS:
Behavioral: My Choice for HIV Prevention (MyChoice) — My Choice for HIV Prevention (MyChoice) is a counselor-delivered shared decision-making approach for pregnant women considering PrEP
  Arms: My Choice for HIV Prevention (MyChoice)
Behavioral: Standard of care (control arm) — Standard of care (control arm) participants will receive comprehensive education on both the advantages and limitations of each PrEP method, including guidance on potential side effects.
  Arms: Standard of care (control arm)

SUMMARY:
Purpose: The overall objective of this pilot study is to evaluate the feasibility, acceptability, and appropriateness of a shared decision-making (SDM) intervention to support personally appropriate decision making about Pre-exposure prophylaxis (PrEP) use during pregnancy and breastfeeding.

Participants: The primary population to be recruited for this study is HIV-negative pregnant women. For qualitative data collection only, investigators will also recruit male partners of these participants, and PrEP counselors and health care workers. The rationale behind focusing on pregnant women is because of the elevated HIV risk faced by women in the perinatal period. Investigators will recruit 50 women to participate in the feasibility pilot study. A subset of these participants will participate in qualitative interviews. Up to 10 male partners and up to 15 study staff will be recruited to participate in qualitative in-depth interviews.

Procedures (methods): Investigators propose a pilot feasibility study of a shared decision making (SDM) intervention for pregnant women considering PrEP. 50 women will be randomized to receive either the SDM intervention addressing daily oral PrEP, Long-acting injectable cabotegravir (CAB-LA), and alternative HIV prevention methods (condoms), or standard of care counselling addressing the same prevention methods. In both studies, investigators will evaluate the feasibility, acceptability, and appropriateness of the intervention and associated study procedures. Women expressing interest in either PrEP method will be referred to government PrEP services.

DETAILED DESCRIPTION:
Study design:

Investigators propose a pilot feasibility study of a shared decision making (SDM) intervention for pregnant women considering PrEP. 50 women will be randomized to receive either the SDM intervention addressing daily oral PrEP, CAB-LA, and alternative HIV prevention methods (condoms), or standard of care counselling addressing the same prevention methods. In both studies, investigators will evaluate the feasibility, acceptability, and appropriateness of the intervention and associated study procedures. Women expressing interest in either PrEP method will be referred to government PrEP services.

Study intervention:

The study intervention, My Choice for HIV Prevention (MyChoice), is a counselor-delivered shared decision-making approach for pregnant women considering PrEP. The intervention counseling will be delivered by trained study staff with a background in psychosocial counseling. The intervention consists of counseling facilitated by a SDM tool. The woman's partner may be present depending on her preference. It begins with a review of HIV risk in pregnancy/breastfeeding including discussion of population-specific risk factors which may apply to the participant. After understanding participant HIV risk and desire for HIV protection, the counselor presents HIV prevention options including CAB-LA, daily oral PrEP, and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (product attributes and personal and interpersonal implications of each method). The counselor reviews information about these valued features for each offered method. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s).

Standard of care (control arm):

Participants randomized to the control arm will PrEP counseling as based on the current standard of care (SOC) . The SOC counseling will be delivered by a trained study staff member. The SOC counselor PrEP counseling according to national guidelines. Per current guidelines, the SOC counseling may include the following elements: An HIV risk assessment according to PrEP eligibility criteria; discussion of a combination prevention approach (PrEP and condoms) and risk reduction strategies. The women will receive comprehensive education on both the advantages and limitations of PrEP, including guidance on managing potential side effects. Subsequently, the counselor will assess the woman's eligibility, willingness, and readiness to start using PrEP. Women choosing oral PrEP during the SOC counseling session will be referred to government services to initiate PrEP. Participants choosing CAB-LA will initiate CAB-LA through the ongoing national pilot program.

Participants will be randomly assigned 1:1 to one of two study arms (intervention or comparison) using permuted block randomization. Participants will be blinded to their assignment, but study staff will not.

Participants choosing oral PrEP during the counselling session in either intervention or comparison arm will receive an assisted referral to government PrEP services at the study site to initiate their selected PrEP method per national guidelines. Participants choosing CAB-LA will initiate CAB-LA through the ongoing national pilot program. No study drug will be administered. Initiation of either PrEP method (i.e., receipt of prescription or injection) will be confirmed through clinic or pharmacy records, as well as information on reasons for non-initiation if applicable.

Investigators plan study follow-up visits at month 1 and month 2 following enrollment. Interviewer-administered questionnaires will be completed at the month 1 follow-up and the final follow-up visit (month 2). Questionnaires will assess study outcomes and associated social and behavioural measures to contextualize understanding of primary study outcomes. A subset of participants will complete in-depth qualitative interviews at month 1. Interviews will provide additional understanding of participant experiences with the intervention and experience using PrEP (if applicable).

ELIGIBILITY:
Inclusion Criteria:

The criteria for pregnant women participants is as follows:

Inclusion criteria

* Age 18 or older
* Documented pregnancy by urine pregnancy test or physical exam
* Documented negative HIV status within the past three months
* Identified factor(s) for elevated risk for HIV acquisition per PrEP national eligibility guidelines
* Willingness to remain in the study site's catchment area over the course of study follow-up and to comply with visit schedule
* Ability and willingness to provide informed consent

Investigators will also conduct interviews with male partners and study staff to assess exploratory qualitative outcomes. All study staff will be eligible to participate in an interview. Male partners will be eligible to participate if they meet the following criteria:

* Referred by a study participant as her romantic partner
* Age 18 or older
* Able and willing to provide informed consent

Exclusion Criteria:

* Positive HIV test at time of screening
* No identified HIV risk factors per national PrEP guidelines
* Risk for intimate partner violence or social harms as a result of participation, in the judgement of the study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure Score | enrollment, final follow up visit (Month 2)
  Intervention acceptability will be defined as the extent to which participants perceive the intervention to be agreeable, palatable, or satisfactory. Acceptability will be assessed through participant self-report using a validated 4-item scale. This scale measures how agreeable and satisfactory women find the intervention (responses rated on a 5-point Likert scale ranging from "Completely Disagree" to "Completely Agree"). Range is 1-5 and higher scores indicate a greater acceptability.
Intervention Appropriateness Measure Score | enrollment, final follow up visit (Month 2)
  Intervention appropriateness will be defined as the perceived relevance and usefulness of the intervention to support decision making about HIV prevention methods. Appropriateness will be assessed through self-report using a validated 4-item scale to measure women's perceptions of its relevance and usefulness (responses rated on a 5-point Likert scale ranging from "Completely Disagree" to "Completely Agree"). Range is 1-5 and higher scores indicate a greater appropriateness.

SECONDARY OUTCOMES:
Mean Number of Women Screened Weekly | At screening
  The number of women screened on a weekly basis will be tracked and an average of weekly screening counts will be taken.
Proportion of Screened Eligible Women Enrolling in the study | At the time of enrollment
  The proportion of women who screen eligible for the study who choose to enroll will be assessed through study records.
Proportion of Enrolled Participants Returning for Follow-Up Visits | 1-month follow-up, 2-month follow-up
  The proportion of enrolled participants who return for 1-month and 2-month follow-up visits will be assessed through study records.
Number of Days Taken to Achieve Enrollment Targets from the Date of Enrollment Initiation | At the time of enrollment
  The total elapsed time in days from the first enrollment to the last will be assessed through study records.
Number of Days Taken to Achieve Retention Targets from the Date of the First Scheduled Follow-up Visit | At the time of enrollment, 2-month follow-up
  The total elapsed time in days from the first enrollment to the last study visit will be assessed through study records.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Hill, PhD,MSPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila Hospital, Lilongwe, Central Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Saidi F, Welch S, Phanga T, Sulpizio C, Paile L, Ngo'ma D, Tsidya M, Chindebvu M, Nkhoma G, Nkhalamba L, Kaliati I, Mkochi N, Chakala H, Kumwenda W, Bula A, Winner P, Munthali T, Nyamaizi A, Keys J, Maman S, Pearce L, Golin C, Chi BH, Hill LM. Supporting Oral and Long-Acting HIV Preexposure Prophylaxis Decision-Making Among Pregnant Women (MyChoice Intervention): Protocol for 2 Pilot Randomized Controlled Trials. JMIR Res Protoc. 2025 Nov 13;14:e76442. doi: 10.2196/76442. PMID 41232107

DOCUMENTS (1):
  • Informed Consent Form (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT06397690/ICF_000.pdf